CLINICAL TRIAL: NCT01146496
Title: A Community Trial to Determine Whether 'Safe Storage' Reduces Pesticide Self-poisoning in Rural Asia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: University of Bristol (Other); University of Oxford (Other); University of Peradeniya (Other); University of Kelaniya (Other); University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Safe Storage Protocol Sep09
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Pesticide Poisoning
Keywords: Pesticide poisoning; Suicide; Unintentional poisoning; Prevention; Cluster randomised controlled trial
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Storage container (Active Comparator): Ultraviolet light resistant plastic in-ground pesticide storage container
  Interventions: Device: Ultraviolet light-resistant plastic in-ground pesticide storage container
- Control (No Intervention)

INTERVENTIONS:
Device: Ultraviolet light-resistant plastic in-ground pesticide storage container — In-ground pesticide storage container to be supplied to every household that uses pesticides in intervention villages
  Arms: Storage container

SUMMARY:
A major global public health priority is to identify effective methods for preventing deaths from pesticide self-poisoning. The aim of this work is to determine whether the provision of lockable storage containers to poor households in rural Asia can reduce the incidence of intentional pesticide self-poisoning. Secondary questions include the effect of these containers on unintentional pesticide poisoning in children and overall self-harm.

DETAILED DESCRIPTION:
We will set up a large community-based, cluster randomised controlled trial of 162 villages (mean adult population 900) in rural Sri Lanka to determine the effectiveness and cost of the provision of safe storage containers to prevent pesticide poisoning.

The study will be based in Anuradhapura District where we have carried out public health studies of pesticide poisoning since 2002. 81 intervention and 81 control villages will be recruited. Randomisation will be clustered, with villages rather than households randomised. A census will be performed at baseline and after 3 years to establish the population demographics and number of person-years exposed.

The primary outcome will be the incidence of pesticide self-poisoning; secondary outcomes will be the incidence of all self-poisoning, all self-harm, fatal self-harm, pesticide poisoning and unintentional paediatric pesticide poisoning. We will use Poisson regression models, taking account of clustering and stratification, for the analysis.

The study will provide definitive evidence concerning the cost-effectiveness of this approach that will determine whether it should be promoted across Asia.

ELIGIBILITY:
Inclusion Criteria:

* Any village in the study area that gives consent to the study

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 223861 (Actual)
Dates: Start 2010-12; Primary Completion 2013-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Eddleston, Principal Investigator — University of Edinburgh; Flemming Konradsen, Study Director — University of Copenhagen
Locations (1):
- Mahaweli H area, Anuradhapura, North Central Province, Sri Lanka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pearson M, Metcalfe C, Jayamanne S, Gunnell D, Weerasinghe M, Pieris R, Priyadarshana C, Knipe DW, Hawton K, Dawson AH, Bandara P, deSilva D, Gawarammana I, Eddleston M, Konradsen F. Effectiveness of household lockable pesticide storage to reduce pesticide self-poisoning in rural Asia: a community-based, cluster-randomised controlled trial. Lancet. 2017 Oct 21;390(10105):1863-1872. doi: 10.1016/S0140-6736(17)31961-X. Epub 2017 Aug 11. PMID 28807536
- [Derived] Knipe DW, Gunnell D, Pieris R, Priyadarshana C, Weerasinghe M, Pearson M, Jayamanne S, Dawson AH, Mohamed F, Gawarammana I, Hawton K, Konradsen F, Eddleston M, Metcalfe C. Is socioeconomic position associated with risk of attempted suicide in rural Sri Lanka? A cross-sectional study of 165 000 individuals. BMJ Open. 2017 Mar 22;7(3):e014006. doi: 10.1136/bmjopen-2016-014006. PMID 28336743
- [Derived] Madsen LB, Eddleston M, Hansen KS, Pearson M, Agampodi S, Jayamanne S, Konradsen F. Cost-effectiveness analyses of self-harm strategies aimed at reducing the mortality of pesticide self-poisonings in Sri Lanka: a study protocol. BMJ Open. 2015 Feb 27;5(2):e007333. doi: 10.1136/bmjopen-2014-007333. PMID 25724984
- [Derived] Pearson M, Konradsen F, Gunnell D, Dawson AH, Pieris R, Weerasinghe M, Knipe DW, Jayamanne S, Metcalfe C, Hawton K, Wickramasinghe AR, Atapattu W, Bandara P, de Silva D, Ranasinghe A, Mohamed F, Buckley NA, Gawarammana I, Eddleston M. A community-based cluster randomised trial of safe storage to reduce pesticide self-poisoning in rural Sri Lanka: study protocol. BMC Public Health. 2011 Nov 21;11:879. doi: 10.1186/1471-2458-11-879. PMID 22104027

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: No intervention
Period: Overall Study
Arm/Group | Storage Container | Control
Started | 114168 | 109693
Completed | 114168 | 109693
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Storage Container | Control | Total
Number analyzed (Participants) | 114168 | 109693 | 223861
Age, Customized [Count of Participants; unit: Participants]
  Number >14 years | 87751 | 84469 | 172220
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Females >14 yrs | 44693 | 43105 | 87798
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Sri Lankan | 114168 | 109693 | 223861
Region of Enrollment [Number; unit: participants]
  Sri Lanka | 114168 | 109693 | 223861

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Pesticide Self-poisoning
Description: Cases identified by survey of local and referral hospitals and by regular interview of primary informants in each village
Time Frame: For three years after intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Storage Container | Control
Number analyzed (Participants) | 114168 | 109693
Participants | 611 | 641

2. Secondary Outcome: Incidence of All Self-poisoning
Description: Cases of self-poisoning identified
Time Frame: For three years post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Storage Container | Control
Number analyzed (Participants) | 114168 | 109693
Participants | 1155 | 1173

3. Secondary Outcome: Incidence of All Self-harm
Time Frame: For three years after intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Storage Container | Control
Number analyzed (Participants) | 114168 | 109693
Participants | 1217 | 1220

4. Secondary Outcome: Incidence of Fatal Self-harm
Time Frame: For three years post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Storage Container | Control
Number analyzed (Participants) | 114168 | 109693
Participants | 82 | 67

5. Secondary Outcome: Incidence of Pesticide Poisoning
Time Frame: For three years post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Storage Container | Control
Number analyzed (Participants) | 114168 | 109693
Participants | 633 | 662

6. Secondary Outcome: Incidence of Unintentional Paediatric Pesticide Poisoning
Time Frame: For three years post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Storage Container | Control
Number analyzed (Participants) | 114168 | 109693
Participants | 18 | 15

ADVERSE EVENTS:
Arm/Group | Storage Container | Control
Serious Adverse Events (participants affected / at risk) | 0/114168 | 0/109693
Other Adverse Events (participants affected / at risk) | 0/114168 | 0/109693

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No